CLINICAL TRIAL: NCT07257419
Title: CD45RA-depleted CD19-CAR T Cell Consolidation After TCR??+ T Cell-depleted Haploidentical Hematopoietic Cell Transplantation for Relapsed/Refractory CD19+ ALL and Lymphoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAPALL; NCI-2025-08364 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Relapsed Pediatric ALL; Hematopoietic Cell Transplantation; Hematologic Malignancy
Keywords: Relapsed/Refractory ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hematologic Neoplasms; Recurrence | interventions — Antilymphocyte Serum; Cyclophosphamide; fludarabine; Thiotepa; Mesna; Melphalan; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- HAPALL Treatment (Experimental): Patients receive a conditioning regimen that will comprise of ATG, Fludarabine, Cyclophosphamide. Melphalan and Thiotepa. Following the conditioning regimen, patients receive infusion of TCRαβ depleted progenitor cell infusion on day 0. Then as early as day + 14 patients will receive the previously manufactured CD19-CAR(Mem) T cell product. Patients will then be monitored for safety and efficacy of the infused CAR T-cell product,
  Cells for infusion are prepared using the CliniMACS system.
  Interventions: Drug: Anti-Thymocyte Globulin (Rabbit); Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Thiotepa; Drug: Mesna; Drug: Melphalan; Drug: Filgrastim; Device: CliniMACS System

INTERVENTIONS:
Drug: Anti-Thymocyte Globulin (Rabbit) — Days -10, -11, -12.
Drug: Cyclophosphamide — 60 mg/kg intravenous once daily on day -9.
Drug: Fludarabine — 30 mg/m2 intravenous once daily for >10 kg, 1 mg/kg intravenous once daily for ≤10 kg on days -4, -5, -6, -7, -8.
Drug: Thiotepa — 5 mg/kg intravenous twice daily on day -3.
Drug: Mesna — Mesna is planned to be administered at 15 mg/kg/dose prior to cyclophosphamide and at approximately 3, 6, and 9 hours after the cyclophosphamide infusion, to give a 1:1 ratio of mesna:cyclophosphamide.
Drug: Melphalan — 70 mg/m2 intravenous once daily for >10 kg, 2.3 mg/kg intravenous once daily for ≤10 kg on days -1, and -2.
Drug: Filgrastim — G-CSF* 10 mcg/kg/day SC days 0, -1, -2, -3, -4, -5.
  Other Names: G-CSF
Device: CliniMACS System — The mechanism of action of the CliniMACS Cell Selection System is based on magnetic-activated cell sorting (MACS). The CliniMACS device is a powerful tool for the isolation of many cell types from heterogeneous cell mixtures, (e.g. apheresis products). These can then be separated in a magnetic field using an immunomagnetic label specific for the cell type of interest.

SUMMARY:
The purpose of this study is to learn more about newer methods of transplanting blood cells donated by a partially matched family member to children with high-risk CD19 positive leukemia ALL.

Primary Objective:

- To assess the safety and feasibility of combining CD19-CAR(Mem) T cells after TCRαβ+ depleted haploidentical donor transplantation for pediatric patients with relapsed/refractory CD19+ B-cell malignancies.

Secondary Objectives:

* To estimate 1-year post-transplant overall survival, relapse free survival, and GVHD-free relapse-free survival (GRFS).
* To estimate cumulative incidence of engraftment, acute and chronic GVHD, and immune-related adverse events, including CRS and ICANS.

DETAILED DESCRIPTION:
This is a Phase I study evaluating the addback of CD19-CAR(Mem) T cells after TCRαβ+ depleted haploidentical donor transplantation for pediatric patients with relapsed/refractory CD19+ B-cell malignancies.

Donors that meet eligibility criteria will be consented to undergo two separate collections: 1) G-CSF mobilized stem cell graft via apheresis for progenitor cell infusion and 2) Non-mobilized peripheral blood mononuclear cells (PBMC) via apheresis for subsequent CAR T-cell manufacturing and DLI if needed.

Patients that meet eligibility criteria to receive therapy will be consented to proceed on study. Treatment will include a conditioning chemotherapy preparative regimen followed by infusion of TCRαβ depleted progenitor cell infusion on day 0. Then as early as day + 14 patients will receive the previously manufactured CD19-CAR(Mem) T cell product. Patients will then be monitored for safety and efficacy of the infused CAR T-cell product, as well as collection of correlative samples.

ELIGIBILITY:
Inclusion Criteria:

Recipient

* Age less than or equal to 21 years
* High risk hematologic malignancy where allogeneic transplantation is the current standard of care. This includes (but is not limited to):

  * High risk CD19+ B cell ALL in CR1 or CR2
  * Any CD19+ B-cell ALL in CR3 or subsequent
* If prior CNS leukemia, it must be treated and in CNS CR
* Left ventricular ejection fraction > 40%, or shortening fraction ≥ 25%
* Creatinine clearance (CrCl) or glomerular filtration rate (GFR) ≥ 50 ml/min/1.73m2
* Forced vital capacity (FVC) ≥ 50% of predicted value; or pulse oximetry ≥ 92% on room air if patient is unable to perform pulmonary function testing
* Karnofsky or Lansky (age dependent) performance score ≥ 50 (See APPENDIX A)
* Bilirubin ≤ 3 times the upper limit of normal for age
* Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) ≤ 5 times the upper limit of normal for age

Donor

* At least single haplotype matched (≥ 4 of 8) family member
* At least 18 years of age
* HIV negative
* Regarding donation eligibility, is identified as either:

  * Completed the process of donor eligibility determination as outlined in 21 CFR 1271 and agency guidance; OR
  * Does not meet 21 CFR 1271 eligibility requirements, but has a declaration of urgent medical need completed by the principal investigator or physician sub-investigator per 21 CFR 1271

Exclusion Criteria:

Recipient

* Has a suitable HLA-identical sibling or suitable 12/12 (HLA-A, B, C, DRB1, DQB1, and DPB1) HLA-matched unrelated donor available in an appropriate time frame
* Any other active malignancy other than the one for which this HCT is indicated
* Received a prior allogeneic HCT at any time
* Received an autologous HCT within the previous 6 months
* Pregnant, if female is of childbearing potential, negative test must be confirmed by serum or urine pregnancy test within 14 days prior to enrollment
* Breast feeding
* Any severe current uncontrolled bacterial, fungal or viral infection

Donor

* Pregnant, negative test must be confirmed by serum or urine pregnancy test within 14 days prior to enrollment if female
* If female, breast feeding

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of combining CD19-CAR(Mem) T cells after TCRαβ+ depleted haploidentical donor transplantation for pediatric patients with relapsed/refractory CD19+ B-cell malignancies. | This will be assessed 100 days post-HCT
  The primary analysis will compute the sample proportions and corresponding binomial exact 95% confidence intervals among evaluable patients for the following toxicities (separately for each toxicity) within 100 days post-HCT: 1) Severe aGVHD defined as Grade 3-4 aGVHD 2) Severe CRS defined as Grade 4 CRS that does not resolve to grade 3 or lower within 72 hours of onset 3) Severe ICANS defined as Grade 4 ICANS that does not resolve to grade 3 or lower within 72 hours of onset 4) TRM defined as death without prior relapse or disease progression within 100 days post-HCT 5) Other toxicity data will also be reported for a complete safety assessment of the study regimen.
To assess the feasibility of combining CD19-CAR(Mem) T cells after TCRαβ+ depleted haploidentical donor transplantation for pediatric patients with relapsed/refractory CD19+ B-cell malignancies. | This will be assessed in the first 60 days post-HCT
  this will be measured by the failure to receive CD19-CAR(Mem) T cells among patients who received HCT. The number of patients who fail to receive addback will be reported as the proportion who were unable to receive addback within 60 days post-HCT

SECONDARY OUTCOMES:
To assess the feasibility of combining CD19-CAR(Mem) T cells after TCRαβ+ depleted haploidentical donor transplantation for pediatric patients with relapsed/refractory CD19+ B-cell malignancies. | This will be assessed in the first 60 days post-HCT
  This will be measured by the failure to receive CD19-CAR(Mem) T cells among patients who received HCT. The number of patients who fail to receive addback will be reported as the proportion who were unable to receive addback within 60 days post-HCT
Estimate 1-year post-transplant relapse free survival | This will be assessed in the first 3 years post-HCT
  This this will be estimated by the Kaplan-Meier method
Estimate cumulative incidence of neutrophil engraftment | This will be assessed in the first 30 days post-HCT
  This will be summarized by cumulative incidence functions estimated by the Kalbfleisch-Prentice method.
Estimate cumulative incidence of platelet engraftment | This will be assessed in the first 100 days post-HCT
  This will be summarized by cumulative incidence functions estimated by the Kalbfleisch-Prentice method.
Estimate cumulative incidence of acute and chronic GVHD | This will be assessed in the first 3 years post-HCT
  This will be summarized by cumulative incidence functions estimated by the Kalbfleisch-Prentice method.
Estimate cumulative incidence of immune-related adverse events | This will be assessed in the first 1 years post-HCT
  This will be summarized by cumulative incidence functions estimated by the Kalbfleisch-Prentice method.

CONTACTS AND LOCATIONS:
Overall Officials: Swati Naik, MBBS, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols